CLINICAL TRIAL: NCT01510795
Title: Impact of a Mineralocorticoid Receptor Antagonist on Chronic Histological Changes in Renal Allograft
Brief Title: Mineralocorticoid Receptor Antagonist and Kidney Allograft Histology
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Clinical Hospital Merkur (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHMN1012
Record Dates: First submitted 2012-01-12; First posted 2012-01-18 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Kidney Failure, Chronic
Keywords: Kidney transplantation; Mineralocorticoid receptors; Spironolactone
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Spironolactone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- retrospective control (No Intervention)
- spironolactone (Active Comparator)
  Interventions: Drug: spironolactone

INTERVENTIONS:
Drug: spironolactone — Spironolactone initiated at 3 months posttransplant at 25 mg qd and up-titrated to 50 mg qd after 14 days. Spironolactone therapy will be maintained for 9 months.
  Other Names: Aldactone
  Arms: spironolactone

SUMMARY:
Chronic allograft nephropathy is one of dominant causes of long term kidney transplant failure. Its main histological determinant is interstitial fibrosis and tubular atrophy. Mechanisms of these changes are multifactorial and are not completely elucidated. Epithelial mesenchymal transition (EMT) might be one of the mechanisms. On molecular level role of renin angiotensin aldosterone system (RAAS) has been recognized. Recently, mineralocorticoid hormone aldosterone has been proposed as a possible direct contributor to the progression of renal injury and fibrosis, beside his well known role as a regulator of extracellular fluid volume and sodium and potassium balance. In this study the investigators will determine the impact of mineralocorticoid receptor antagonist use on progression of chronic scores in transplanted kidney over one year. The investigators hypothesis is that spironolactone use in kidney transplant patients will slow down progression of chronic histological changes- interstitial fibrosis, tubular atrophy and arteriolar hyalinosis.

DETAILED DESCRIPTION:
Chronic allograft nephropathy (CAN) is the main cause of long term kidney transplant failure. Its main histological determinant is interstitial fibrosis and tubular atrophy, but mechanisms of these changes are not completely elucidated and seem to be multifactorial. It seems that these histological changes develop as a consequence of immunological and non-immunological mechanisms. Study from Nankivell and al. defined two phases of CAN, early, attributed to immunological mechanisms; acute rejection, persistent subclinical rejection and ischemic- reperfusion injury, and late injury, characterized with progressive arteriolar hyalinosis, glomerulosclerosis andInterstitial fibrosis and tubular atrophy (IF/TA), which was attributed in part to calcineurin inhibitor use and in part to ongoing immunologic injury.

In vitro studies and animal studies have shown epithelial mesenchimal transition as one of possible mechanisms and early markers of subsequent IF/TA. EMT is defined as process where completely differentiated epithelial cells undergo transition into fibroblast phenotype cells.

It is known that on molecular level RAAS has crucial role in development of progressive renal injury and fibrosis. Role of angiotensin II in progression of chronic kidney injury is established and well known. It mediates kidney injury by increasing intraglomerular capillary pressure leading to ultrafiltration of plasma proteins and by promoting cell growth and fibroproliferative effects.

It is hypothesized that aldosterone as a component of RAAS may also have direct role in proinflammatory and profibrotic mechanisms of initiation and progression of kidney injury. Aldosterone is a mineralocorticoid hormone produced in adrenal cortex zona glomerulosa and has crucial role as a regulator of extracellular fluid volume and sodium and potassium balance.

It has been shown in the rat models that aldosterone activates mTOR kinase, which promotes cell proliferation and contributes in early phases of injury healing. However, a prolonged activation of mTOR seems to promote development of interstitial fibrosis.

Although the molecular pathways of aldosterone-mediated renal injury have not yet been fully elucidated, aldosterone may directly contribute to the final common pathway of renal fibrosis. In vitro studies have shown that aldosterone significantly increases TGF beta and fibronectin production by mesangial cells in culture and that this event is abolished by the aldosterone antagonist spironolactone. Randomized studies have shown beneficial role of blockade of mineralocorticoid receptors in heart failure. Also studies have shown beneficial role of mineralocorticoid receptor blockade with nonselective antagonist spironolactone in reducing albuminuria in both diabetic and non diabetic chronic kidney disease (CKD) and antiproteinuric effect of a selective aldosterone inhibitor, eplerenone in type 2 diabetic patients with microalbuminuria. Role of mineralocorticoid receptor blockade in kidney transplant recipients has not been extensively evaluated so far.

In this study we hypothesized that use of a mineralocorticoid receptor antagonist, spironolactone, may contribute to slower progression of chronic histological changes in renal allografts.

ELIGIBILITY:
Inclusion Criteria:

* kidney and kidney-pancreas recipients, including patients with delayed graft function ( DGF). DGF will be defined as the dialysis need in first 7 days after transplantation

Exclusion Criteria:

1. Baseline plasma potassium level above 5.1 µmol/L
2. Patients on ACE inhibitor or ARB-s therapy
3. Patients with eGFR < 30 ml/min (estimated by MDRD formula)
4. Patents younger than 18 yr
5. Patients with hypersensitivity to spironolacton

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-06 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Difference in 6-month changes in chronic Banff scores between spironolactone and retrospective control group | 6 months

SECONDARY OUTCOMES:
Difference in chronic Banff scores between spironolactone and retrospective control group at 12 months, eGFR at 6 and 12 months, urinary protein/creatinine ratio and urinary albumin/creatinine ratio at 6 and 12 months | 6-12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bojana Maksimović, MD, Principal Investigator — Clinical Hospital Merkur; Mladen Knotek, MD, PhD, Study Director — Clinical Hospital Merkur